CLINICAL TRIAL: NCT01766505
Title: Randomized, Open-label, Phase 4 Study to Evaluate Efficacy and Safety of Candesartan and Losartan in the Patients With Hypertension and Heart Failure.
Brief Title: The Study to Evaluate Efficacy and Safety of Candesartan vs Losartan in Hypertension With Heart Failure (HONOR)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of the subjects
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: m111HHF11F
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Hypertension
Keywords: hypertension, heart failure, candesartan, losartan
MeSH Terms: conditions — Hypertension; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Candemore tablet (Experimental): Candemore tablet: candesartan cilexetil 8mg, 16mg, 32mg/tab, orally, 1 tablet once a day during 16 weeks
  Interventions: Drug: Candemore tablet
- Cozzar tablet (Active Comparator): Cozzar tablet: Losartan potassium 50mg, 100mg/cap, orally, 1 capsule once a day during 16 weeks
  Interventions: Drug: Cozzar tablet

INTERVENTIONS:
Drug: Candemore tablet — Candemore tablet 8, 16, or 32mg/tab, per oral, a tablet once a day during 16 weeks.
  dosage is depends on the sitting blood pressure.
  Arms: Candemore tablet
Drug: Cozzar tablet — Cozzar tablet: 8mg, 16mg, 32mg/tablet, per oral, a tablet a day during 16 weeks dosage depends on sitting blood pressure
  Arms: Cozzar tablet

SUMMARY:
The purpose of this study is to compare efficacy and safety of candesartan and losartan in hypertension with heart failure.

DETAILED DESCRIPTION:
This is a randomized, open-label, phase 4 study. wash out periods need at least 14 days if the patients take ARB or ACE inhibitor to control Blood pressure. Patients take Candemore or Cozzar once a day during 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients who aged above 19 and below 75
* Patients with 90~109mmHg average sitting DBP on baseline
* NYHA class 2~4
* Patients who agreement with written informed consent

Exclusion Criteria:

* above 110mmHg sitting DBP and/or 180mmHg sitting SBP
* Patients who have difference values that above 20mmHg sitting SBP or 10mmHg sitting DBP in both arms on screening
* Patients who have medical history that secondary hypertension or rule out secondary hypertension
* malignant hypertension
* symptomatic postural hypotension
* right heart failure due to pulmonary disease
* etc.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
change from baseline average sitting DBP(diastolic blood pressure)at 16 weeks | baseline, 16 weeks

SECONDARY OUTCOMES:
change from baseline average sitting DBP(diastolic blood pressure)at 8 weeks | baseline, 8 weeks
change from baseline average sitting SBP(systolic blood pressure)at 8 weeks | baseline, 8 weeks
change from baseline average sitting SBP(systolic blood pressure)at 16 weeks | baseline, 16 weeks
ratio of normalize from baseline blood pressure at 16 weeks | baseline, 16 weeks
  normalize means that sitting SBP and DBP is below 140mmHg and 90mmHg
response ratio from baseline blood pressure at 16 weeks | baseline, 16 weeks
  response means that decrease in sitting DBP and SBP is above 10mmHg and 20mmHg
change from baseline LVEF(left ventricular ejection fraction at 16 weeks | baseline, 16 weeks
change from baseline LVEDD(left ventricular end-diastolic diameter)at 16 weeks | baseline, 16 weeks
change from baseline LV(left ventricular) mass at 16 weeks | baseline, 16 weeks
change from baseline PWV(pulse wave velocity) mass at 16 weeks | baseline, 16 weeks

OTHER OUTCOMES:
rate of adverse event | up to 16 weeks
medication history | up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Myungho Jeong, phD, Principal Investigator — Chonnam National University Hospital
Locations (9):
- South Korea (9):
  - Chungnam national university hospital, Daejeon
  - The catholic university of Korea, Daejeon st. Mary's Hospital, Daejeon
  - Konyang university hospital, Daejeon
  - Eulji University Hospital, Daejeon
  - Chunnam National University Hospital, Gwangju
  - Kwangju Christian Hospital, Gwangju
  - Presbyterian Medical Center, Jeonju
  - Chunbuk National University Hospital, Jeonju
  - ST.Carollo hospital, Suncheon